CLINICAL TRIAL: NCT00385307
Title: An Eight-Week, Double-Blind, Placebo-Controlled, Multicenter Study With Paroxetine (10 mg qd) as Positive Control, Evaluating the Efficacy, Safety, Tolerability of Two Fixed Doses of SR58611A (175 mg q12/ 350 mg q12) in Outpatients With MDD
Brief Title: Efficacy and Safety of SR58611A in Patients With Major Depressive Disorder (SIRIUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6607
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Clinical Trials; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — amibegron; Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: amibegron (SR58611A)

SUMMARY:
To evaluate the efficacy of two fixed doses of SR58611A (175 mg q12 and 350 mg q12) compared to placebo in patients with Major Depressive Disorder (MDD) using paroxetine (20 mg qd) as positive control. In addition, the tolerability and safety of SR58611A in patients with MDD will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Major Depressive Disorder diagnosed according to Diagnostic and Statistical Manual of Mental Disorders DSM-IV-TR
* Patient meets criteria for a recurrent Major Depressive Episode (MDE)
* Patient meets severity assessments of depression specified by the study

Exclusion Criteria:

* Patient is at immediate risk for suicidal behavior
* Patient is with a unstable medical condition
* Patient with psychotic features, catatonic features, seasonal pattern or postpartum onset
* Patient has taken concomitant treatment that may interfere with valid collection or interpretation of study data
* Patient has been treated with non-pharmacologic therapy intended to treat depression in the past 6 months
* Patient has been treated with paroxetine (Paxil) within the previous 6 months
* Patient is pregnant or breastfeeding, or likely to become pregnant during the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total score of a depression rating scale at 8 weeks

SECONDARY OUTCOMES:
Safety assessments

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States